CLINICAL TRIAL: NCT01043679
Title: A Randomized Open-label Active-controlled Study to Evaluate the Efficacy and Safety of Utapine Versus Seroquel in Patients With Bipolar Mania
Brief Title: Efficacy and Safety of Utapine vs. Seroquel in Patients With Bipolar Mania
Acronym: UtapMani
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: IRB TCVGH, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01122009/S09070
Record Dates: First submitted 2010-01-06; First posted 2010-01-07 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Bipolar, Mania; Utapine; Seroquel
Keywords: Bipolar, Mania; Utapine; Seroquel
MeSH Terms: conditions — Mania | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Seroquel (Active Comparator): Efficacy and Safety of Seroquel
  Interventions: Drug: Seroquel
- Utapine (Active Comparator): Efficacy and Safety of Utapine
  Interventions: Drug: Utapine

INTERVENTIONS:
Drug: Utapine — Efficacy and Safety of Utapine
  Arms: Utapine
Drug: Seroquel — Efficacy and Safety of Seroquel
  Arms: Seroquel

SUMMARY:
The goal of this research is to evaluate the safety as well as effectiveness of Utapine and Seroquel in bipolar I disorder patients.

DETAILED DESCRIPTION:
Utapine and Serquel belong to anti-bipolar medication family, both are approved by DOH (Department of Health, Taiwan), both has same ingredient but different manufacture. From clinical trial reports, both has excellent effectiveness and safety. The goal of this research is to evaluate the safety as well as effectiveness of Utapine and Seroquel in bipolar I disorder patients for different ingredient and different manufacture.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18-65 years with diagnosis of bipolar I disorder who will be included by DSM-IV criteria made at least one manic or mixepisode record before study entry.
2. Having a minimum score of 20 on the Young Mania Rating Scale (YMRS), plus a score of at least 4 on two of the core YMRS items of Irritability,Speech, Content, and Disruptive/Aggressive Behavior.
3. At least 4 will be on the Severity of Illness item of the Clinical Global ImpressionsNBipolar(CGINBP)assessment tool.
4. Patient with good compliance to study medicine and adherence to study protocol.

Exclusion Criteria:

1. Had received treatment with clozapine within 28 days of the start of the trial.
2. Had been hospitalised for 3 weeks or longer for the index manic episode.
3. DSM-IV criteria for rapid cycling or a current mixed episode.
4. Intolerance or lack of response to quetiapine or clozapine before this trial be diagnosed by investigator.
5. Neurodegenerative disease eg:Parkinson desease、Huntington disease、Pick's disease.
6. Medicine or drugs which can change mental condition be judged by investigator.
7. EKG abnormality
8. Drug or alcohol abuser

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Hong Chan, MD.,MS., Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan